CLINICAL TRIAL: NCT04550052
Title: A-SPIRE Heart Failure: Utilizing Physiologic Information From Spire Health Tags to Identify Heart Failure Patients At-Risk for Hospital Readmission: A Pilot Feasibility Study
Brief Title: A-SPIRE Heart Failure: Utilizing Health Tags to Identify Patients at Risk for Hospital Readmissions
Acronym: A-SPIRE-HF
Status: Active, not recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Spire, Inc. (Industry)
Responsible Party: Principal Investigator, Valentina Kutyifa, Associate Professor of Medicine (Cardiology), University of Rochester
Other Study IDs: 00004060
Record Dates: First submitted 2020-08-27; First posted 2020-09-16 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
Keywords: Spire Health Tag
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the use of the Spire Health Tags in heart failure patients to determine the feasibility of capturing signals of respiration, pulse rate, activity, sleep patterns, and stress levels following HF hospitalization.

DETAILED DESCRIPTION:
Over 5 million Americans suffer from heart failure (HF), and treating HF as a chronic condition is associated with significant costs. In addition, about 24% of the patients discharged with a primary diagnosis of HF are readmitted to the hospital within 30 days, representing a significant public health burden. While there have been efforts to predict and reduce 30-day hospital readmission initiated by the Centers for Medicare and Medicaid Services (CMS), no studies utilized daily physiologic data from wearables to identify at-risk patients.

The overall goal of this proposed pilot feasibility study is to utilize the Spire Health Tags in a heart failure patient population to ascertain the feasibility of capturing appropriate signals of respiration, pulse rate, activity, sleep patterns, and stress levels (calm/focused/tense during the day) for > 80% of the time in patients following HF hospitalization for a 30-day period. The investigators will do exploratory analysis of the changes in these physiologic variables during a 30-day period following HF hospitalization to identify risk markers that could predict 30-day readmission.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age or older;
* Admitted for acute heart failure;
* Expected to be discharged from hospitalization;
* Able to give consent;
* Willing to use the Spire Health Tags for 30 days continuously.

Exclusion Criteria:

* Unable or unwilling to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients discharged following heart failure hospitalization,
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To ascertain the feasibility of capturing appropriate signals of pulse rate for > 80% of the time in patients following HF hospitalization for a 30-day period. | 30 Days
  We will evaluate capturing data in at least 80% of the time (24 days of the 30 days) using the Spire Health Tags during a 30 day period.
To ascertain the feasibility of capturing appropriate signals of activity for > 80% of the time in patients following HF hospitalization for a 30-day period. | 30 Days
  We will evaluate capturing data in at least 80% of the time (24 days of the 30 days) using the Spire Health Tags during a 30 day period.
To ascertain the feasibility of capturing appropriate signals of sleep patterns for > 80% of the time in patients following HF hospitalization for a 30-day period. | 30 Days
  We will evaluate capturing data in at least 80% of the time (24 days of the 30 days) using the Spire Health Tags during a 30 day period.
To ascertain the feasibility of capturing appropriate signals of stress levels (calm/focused/tense during the day) for > 80% of the time in patients following HF hospitalization for a 30-day period. | 30 Days
  We will evaluate capturing data in at least 80% of the time (24 days of the 30 days) using the Spire Health Tags during a 30 day period.

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Kutyifa, MD, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):399-410. doi: 10.1161/01.cir.0000442015.53336.12. No abstract available. PMID 24446411
- [Result] Keenan PS, Normand SL, Lin Z, Drye EE, Bhat KR, Ross JS, Schuur JD, Stauffer BD, Bernheim SM, Epstein AJ, Wang Y, Herrin J, Chen J, Federer JJ, Mattera JA, Wang Y, Krumholz HM. An administrative claims measure suitable for profiling hospital performance on the basis of 30-day all-cause readmission rates among patients with heart failure. Circ Cardiovasc Qual Outcomes. 2008 Sep;1(1):29-37. doi: 10.1161/CIRCOUTCOMES.108.802686. PMID 20031785
- [Result] Dharmarajan K, Hsieh AF, Lin Z, Bueno H, Ross JS, Horwitz LI, Barreto-Filho JA, Kim N, Bernheim SM, Suter LG, Drye EE, Krumholz HM. Diagnoses and timing of 30-day readmissions after hospitalization for heart failure, acute myocardial infarction, or pneumonia. JAMA. 2013 Jan 23;309(4):355-63. doi: 10.1001/jama.2012.216476. PMID 23340637
- [Result] Amarasingham R, Patel PC, Toto K, Nelson LL, Swanson TS, Moore BJ, Xie B, Zhang S, Alvarez KS, Ma Y, Drazner MH, Kollipara U, Halm EA. Allocating scarce resources in real-time to reduce heart failure readmissions: a prospective, controlled study. BMJ Qual Saf. 2013 Dec;22(12):998-1005. doi: 10.1136/bmjqs-2013-001901. Epub 2013 Jul 31. PMID 23904506
- [Result] Fang J, Wylie-Rosett J, Cohen HW, Kaplan RC, Alderman MH. Exercise, body mass index, caloric intake, and cardiovascular mortality. Am J Prev Med. 2003 Nov;25(4):283-9. doi: 10.1016/s0749-3797(03)00207-1. PMID 14580628
- [Result] Seefeldt V, Malina RM, Clark MA. Factors affecting levels of physical activity in adults. Sports Med. 2002;32(3):143-68. doi: 10.2165/00007256-200232030-00001. PMID 11839079